CLINICAL TRIAL: NCT07377682
Title: Observational Prospective Study in Patients With Major Depressive Disorder and Mild Cognition Impairment Treated With Trazodone in a Real-world Setting (TRACOMDD)
Brief Title: Real-world Clinical Response to Trazodone in Italy, Poland, and Romania
Status: Recruiting | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: IQVIA Solutions (Unknown)
Responsible Party: Sponsor
Other Study IDs: 039(Z)MD24063
Record Dates: First submitted 2025-12-17; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Cognition Disorders in Old Age
Keywords: Depression; Major Depressive Disorder; Cognition
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TRACOMDD study is a study with the intention to describe the real-world use of trazodone and the clinical response in a sub-group of patients affected by Major Depressive Disorder and Mild Cognitive impairment, by collecting data from standard clinical practice in Italy, Poland, and Romania

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 55 or older.
* Patients who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for MDD diagnosis.
* Patients experiencing a current major depressive episode of at least moderate severity, defined by a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≥20 at enrolment.
* Patients with a diagnosis of MCI (also referred to as "mild neurocognitive disorder") according to the DSM-5 criteria.
* Patients who start treatment with trazodone hydrochloride (prolonged release) with starting dosage according to SmPC at enrolment visit (or at latest within one week).
* Patients legally capable of giving their written consent to participate in the study (including personal data processing) and willing to comply with all study procedures as per clinical judgement.

Exclusion Criteria:

* Patients who meet any of the contraindications to the administration of trazodone according to the approved local SmPC.
* Known hypersensitivity or allergy to the active ingredient and/or to any component of the study medication.
* Concomitant treatment with other antidepressant drugs, mood stabilizers, antipsychotics, and/or proved resistance to trazodone monotherapy.
* Patients with current diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, severe personality disorder, mental retardation, organic mental disorders, or mental disorders due to a general medical condition.
* Patients with previous or current history of any neurological condition that, in the opinion of the Investigator, might compromise participation in the study.
* Patients participating in any interventional study in the 30 days prior to the enrolment visit.
* Patients with ongoing pregnancy or breast-feeding at enrolment visit.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Major Depressive Disorder and mild cognition impairment treated with trazodone
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms severity (MADRS) | At 24 weeks from treatment
  To describe the response in terms of depressive symptoms severity (as measured by Montgomery-Åsberg Depression Rating Scale [MADRS]) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a widely used clinician-rated scale designed to measure the overall severity of core symptoms of depression in patients with MDD.
  It consists of 10 items: nine of the items are based upon patient report and one is on the rater's observation during the rating interview.
  MADRS items are rated on a 7-point scale, where 0 refers to the lack of the symptom and 6 refers to the most severe level of the symptom.
  The total score is the sum of the items and ranges from 0 to 60, with higher scores indicating greater severity of depressive symptoms.
  The MADRS is completed by the Investigator at each scheduled visit and the results will be entered into the eCRF.

SECONDARY OUTCOMES:
Depressive symptoms severity (MADRS) | At 12 weeks from treatment
  To describe the response in terms of depressive symptoms severity (as measured by MADRS) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The Montgomery-Åsberg Depression Rating Scale (MADRS) is a widely used clinician-rated scale designed to measure the overall severity of core symptoms of depression in patients with MDD.
  It consists of 10 items: nine of the items are based upon patient report and one is on the rater's observation during the rating interview.
  MADRS items are rated on a 7-point scale, where 0 refers to the lack of the symptom and 6 refers to the most severe level of the symptom.
  The total score is the sum of the items and ranges from 0 to 60, with higher scores indicating greater severity of depressive symptoms.
  The MADRS will be completed by the Investigator at each scheduled visit and the results will be entered into the eCRF.
Clinical response (CGI) | At 24 weeks from treatment
  To describe the clinical response (as measured by Clinical Global Impression [CGI]) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The Clinical Global Impression (CGI) is a 3-item clinician-rated scale that measures the severity of psychopathology (CGI-S), the global improvement of the patient (CGI-I) and therapeutic response (CGI-E). CGI-S and CGI-I are rated on a 7-point scale.
  For CGI-S, a score of 1 indicates lack of illness and 7 indicates the greatest severity.
  For CGI-I, the score ranges from 1, referring to the biggest improvement, to 7, referring to the biggest worsening. CGI-E evaluates 2 dimensions of the therapeutic response, namely, the therapeutic effect and side effects, rated on 4 levels.
  The assessment is performed on a 4x4 scale, with scores ranging from 1 to 16. The CGI will be completed by the Investigator at V1 (only CGI-S) and V3 (or early termination visit) and the results will be entered into the eCRF
Cognitive functioning (MoCA) | At 24 weeks from treatment
  To describe the response in terms of cognitive functioning (as measured by Montreal Cognitive Assessment [MoCA] and Repeatable Battery for the Assessment of Neuropsychological Status [RBANS]) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The Montreal Cognitive Assessment (MoCA) is a brief screening tool which includes 11 tasks assessing several cognitive domains, namely, memory, visuospatial abilities, executive functions, attention, concentration, language, and orientation to time and place. The total score ranges from 0 to 30.
  A score of 26 or above is considered normal, while scores below 26 indicate potential mild cognitive impairment or more serious.
  In addition, a correction for education is applied by adding 1 point for subjects with less than 12 years of education. The MoCA will be administered to the patient by the Investigator at V1 and V3 (or early termination visit) and the results will be entered into the eCRF.
Sleep quality (SQS) | At 24 weeks from treatment
  To describe the response in terms of sleep quality (as measured by the single-item Sleep Quality Scale [SQS]) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The Sleep Quality Scale (SQS) is a single-item validated questionnaire evaluating overall quality of sleep using a visual analogue scale (VAS), with values ranging from 0 (terrible) to 10 (excellent).
  The recall period for the scale is seven days. The SQS is completed by the patient at V1 and V3 (or early termination visit) and the results will be and entered into the eCRF by the Investigator.
To describe the response in terms of quality of life (EQ-5D-5L) | At 24 weeks from treatment
  To describe the response in terms of quality of life (as measured by the Euro-Quality of Life 5 dimensions - 5 level [EQ-5D-5L]) start among patients with moderate-severe MDD and with MCI treated with prolonged release trazodone.
  The EuroQol-5 Dimensions - 5 Levels (EQ-5D-5L) is a brief and generic tool to measure patient-reported health status.
  It consists of two parts. EQ-5D-5L includes 5 questions covering 5 domains of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression).
  Each question is rated on 5 levels of response, ranging from no problems to extreme problems. The measure also includes a visual analogue scale (EQ-VAS) which requires patients to rate their own health from 0 to 100,representing, respectively, the worst and best imaginable health status.
  The EQ-5D-5L will be completed by the patient at V1 and V3 (or early termination visit) and the results will be entered into the eCRF by the Investigator.
Absolute and relative frequency of patients | Over 24 weeks
  Analyze the response absolute and relative frequency of patients with moderate-severe MDD and with MCI discontinuing trazodone during the study period and reasons for discontinuation.
  Analyze the response absolute and relative frequency of patients with moderate-severe MDD and with MCI starting another anti-depressant during the study period and type of anti-depressant.
  Analyze the response absolute and relative frequency of concomitant medications.
Serious adverse events of prolonged release trazodone | Over 24 weeks
  Analyze the absolute and relative frequency of patients experiencing serious adverse events.
  Descriptive statistics will be provided for details of AEs, such as severity, outcome, seriousness, causality, and action taken.
  AEs will be coded using the MedDRA.
Drug related adverse events of prolonged release trazodone | Over 24 weeks
  Analyze absolute and relative frequency of patients experiencing drug related adverse events.
  Descriptive statistics will be provided for details of AEs, such as severity, outcome, seriousness, causality, and action taken.
  AEs will be coded using the MedDRA.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, Principal Investigator — CAMPUS BioMedico
Locations (1):
- Poradnia Medycyna Miłorząb: pl. Pokoju 3/4, 90-227 Łódź. Poland, Lodz, Poland, Poland